CLINICAL TRIAL: NCT05143047
Title: Development and Evaluation of a Health Literacy-Informed Communication Intervention for Discharge Medication Counseling in Hospitalized Children
Brief Title: Discharge Medication Counseling in Hospitalized Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Principal Investigator, Alison Carroll, Clinical Instructor in Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 8194
Record Dates: First submitted 2021-11-19; First posted 2021-12-03 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-03

CONDITIONS: Medication Management

STUDY DESIGN:
Intervention Model Description: Participants are randomized to control or intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in the usual care group will receive standard-of-care discharge communications per unit routine, including counseling regarding prescribed medications and post-discharge instructions, return precautions, and follow-up appointments by the pediatric nursing staff.
- Intervention (Experimental): Participants in the intervention group will receive supplementary medication discharge instructions in addition to the standard communications. They will receive instructions on how to submit information and complete study surveys securely through their cellphones during their child's home treatment period.
  Interventions: Behavioral: Medication counseling

INTERVENTIONS:
Behavioral: Medication counseling — Participants will receive a customized written medication instruction sheet which includes a picture of an oral dosing syringe indicating the patient's dose as well as a chart showing medication name, dose, route, frequency, duration, next dose due, side effects, and storage information. In addition, participants will be shown how to draw up their child's dose using an oral syringe and then will be asked to practice this task ("show-back"). "Teach-back" will be used to ensure participant's understanding of medication details.
  Arms: Intervention

SUMMARY:
Our objective is to design and test the efficacy of a health-literacy-informed discharge medication counseling intervention in the inpatient setting to reduce medication dosing errors and improve adherence in hospitalized children discharged on a new liquid medication.

DETAILED DESCRIPTION:
The goal of this research is to improve discharge medication adherence and reduce medication dosing errors following pediatric hospitalization. Medication errors are one of the most common healthcare-associated adverse events in pediatrics, with approximately one out-of-hospital medication error occurring every 8 minutes among children < 6 years of age. Liquid medications account for the majority of pediatric dosing errors which is likely due to liquid medications' inherent dosing complexities, including the need for weight-based dosing, different concentrations of medications, and parental use of unstandardized dosing instruments. The increased stress and exhaustion that many caregivers experience during a hospitalization, coupled with the need to assimilate large amounts of information pertaining to post-discharge care, makes transitioning to home from an inpatient stay a particularly high risk period for medication errors. Communication challenges, particularly failure to consider caregiver health literacy, further compounds the risk for medication errors due to poor caregiver comprehension and adherence to discharge instructions.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of children up to 6 years old who are hospitalized on a general inpatient hospital medicine teams
* Caregivers must speak English or Spanish
* Participants' children must be discharged home on new scheduled liquid medication for minimum 3 days.

Exclusion Criteria:

* Medication will be administered by home health nurse
* Child is in state/protected custody
* Medication prescription is prescribed to pharmacy other than hospital outpatient pharmacy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Carroll, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Monroe Carell Jr. Children's Hospital - Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carroll AR, Johnson JA, Stassun JC, Greevy RA, Mixon AS, Williams DJ. Health Literacy-Informed Communication to Reduce Discharge Medication Errors in Hospitalized Children: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2350969. doi: 10.1001/jamanetworkopen.2023.50969. PMID 38227315

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Participants (caregivers) in the usual care group will receive standard-of-care discharge communications per unit routine, including counseling regarding prescribed medications and post-discharge instructions, return precautions, and follow-up appointments by the pediatric nursing staff.
- Intervention: Participants (caregivers) in the intervention group will receive supplementary medication discharge instructions in addition to the standard communications. They will receive instructions on how to submit information and complete study surveys securely through their cellphones during their child's home treatment period.
  Medication counseling: Participants will receive a customized written medication instruction sheet which includes a picture of an oral dosing syringe indicating the patient's dose as well as a chart showing medication name, dose, route, frequency, duration, next dose due, side effects, and storage information. In addition, participants will be shown how to draw up their child's dose using an oral syringe and then will be asked to practice this task ("show-back"). "Teach-back" will be used to ensure participant's understanding of medication details.
Period: Overall Study
Arm/Group | Control | Intervention
Started | 99 | 99
Completed | 72 | 79
Not Completed | 27 | 20

BASELINE CHARACTERISTICS:
Population: Participants in this study are the caregivers of children discharged from the hospital. The children themselves are not enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 99 | 99 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.4 (2.0) | 2.4 (2.1) | 2.4 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 43 | 88
  Male | 54 | 56 | 110
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Black/African American | 16 | 10 | 26
  White | 67 | 75 | 142
  More than one race | 12 | 9 | 21
  Prefer not to answer | 3 | 1 | 4
  Hispanic/Latino ethnicity | 25 | 19 | 44
Uses medication(s) regularly [Count of Participants; unit: Participants] | 24 | 26 | 50
2+ hospitalizations in last year [Count of Participants; unit: Participants] | 19 | 14 | 33
Complex chronic condition present [Count of Participants; unit: Participants] | 20 | 27 | 47
Payer [Count of Participants; unit: Participants]
  Government | 72 | 52 | 124
  Private | 26 | 46 | 72
  No insurance | 0 | 1 | 1
  Other | 1 | 0 | 1
Discharge medication type [Count of Participants; unit: Participants]
  Antimicrobials | 85 | 85 | 170
  Anticonvulsants | 2 | 2 | 4
  Steroids | 4 | 2 | 6
  Gastrointestinal agents/antacids | 3 | 4 | 7
  Other medications | 5 | 6 | 11
Caregiver age [Mean (Standard Deviation); unit: years] | 30.6 (5.9) | 32.1 (7.0) | 31.4 (6.5)
Cargiver sex [Count of Participants; unit: Participants]
  male | 5 | 7 | 12
  female | 94 | 92 | 186
Caregiver relationship to child [Count of Participants; unit: Participants]
  mother | 91 | 91 | 182
  father | 7 | 7 | 14
  grandmother | 1 | 0 | 1
  legal guardian | 0 | 1 | 1
Caregiver race [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Black/African American | 15 | 13 | 28
  Native Hawaiian/Pacific Islander | 0 | 3 | 3
  White | 78 | 80 | 158
  More than one race | 2 | 1 | 3
  Prefer not to answer | 4 | 1 | 5
Caregiver Hispanic/Latino [Count of Participants; unit: Participants] | 24 | 12 | 36
Caregiver language [Count of Participants; unit: Participants]
  English | 80 | 91 | 171
  Spanish | 19 | 8 | 27
Caregiver born outside of U.S. [Count of Participants; unit: Participants] | 26 | 14 | 40
Caregiver education [Count of Participants; unit: Participants]
  Less than high school diploma | 16 | 14 | 30
  High school degree or equivalent | 31 | 23 | 54
  Some college, no degree | 28 | 30 | 58
  College degree | 16 | 22 | 38
  Graduate degree | 8 | 10 | 18
Caregiver difficulty paying bills at home [Count of Participants; unit: Participants] | 21 | 14 | 35
Caregiver Newest Vital Sign score (max=6) [Count of Participants; unit: Participants] — The Newest Vital Sign is a validated screening tool that identifies those at risk for low health literacy. [Weiss BD et al; Ann Fam Med. 2005 Nov-Dec;3(6):514-22.] Caregivers were given the three-minute screening test at the time of enrollment.
  Participants
    Low Health Literacy (score = 0-1) | 15 | 11 | 26
    Marginal Health Literacy (score = 2-3) | 42 | 31 | 73
    Adequate Health Literacy (score = 4-6) | 42 | 57 | 99

OUTCOME MEASURES:

1. Primary Outcome: Observed Dosing Accuracy
Description: Participants (caregivers) will be asked to draw up a dose of their child's liquid medication using the provided oral dosing syringe and send a secure picture of the syringe via myCap (secure phone application designed to collect patient-centered outcomes for research studies) to research study staff. The primary outcome will be assessed as a continuous percent difference from the prescribed dose (in milliliters) documented in the electronic health record. Study staff assessing amount in picture are blinded to group assignment.
Time Frame: During follow-up survey assessment 48-72 hours following hospital discharge
Population: Number of participants analyzed represent those enrolled and randomized minus those withdrawn or lost to follow-up.
Measure: Mean (Standard Deviation); unit: percent difference
Arm/Group | Control | Intervention
Number analyzed (Participants) | 72 | 79
percent difference | 3.3 (5.1) | 1.0 (2.2)
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Reported Dosing Accuracy
Description: Participants (caregivers) will be asked to report the prescribed volume (in milliliters) of medication to be given with each dose during the follow-up myCap survey. This will be compared to the prescribed dose in the electronic medical record.
Time Frame: During follow-up survey assessment 48-72 hours following hospital discharge
Population: Number of participants analyzed represent those enrolled and randomized minus those withdrawn or lost to follow-up.
Measure: Mean (Standard Deviation); unit: percent difference
Arm/Group | Control | Intervention
Number analyzed (Participants) | 68 | 75
percent difference | 2.0 (6.0) | 0.4 (3.0)
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.04, t-test, 2 sided

3. Secondary Outcome: Correct Medication Name
Description: Participants (caregivers) will be asked in a follow-up survey to provide the name of their child's discharge medication. This will be scored as correct if it matches the name of the medication prescribed in the electronic health record.
Time Frame: During follow-up survey assessment 48-72 hours following hospital discharge
Population: Number of participants analyzed represent those enrolled and randomized minus those withdrawn or lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 69 | 76
Participants | 60 | 70
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.42, Fisher Exact

4. Secondary Outcome: Correct Medication Indication
Description: Participants (caregivers) will be asked in a follow-up survey to provide the indication for their child's discharge medication. This will be scored as correct if it matches the indication for the medication prescribed in the electronic health record.
Time Frame: During follow-up survey assessment 48-72 hours following hospital discharge
Population: Number of participants analyzed represent those enrolled and randomized minus those withdrawn or lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 69 | 76
Participants | 59 | 71
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.17, Fisher Exact

5. Secondary Outcome: Correct Medication Dose
Description: Participants (caregivers) will be asked in a follow-up survey to provide the dosage for their child's discharge medication. This will be scored as correct if it matches the indication for the medication prescribed in the electronic health record.
Time Frame: During follow-up survey assessment 48-72 hours following hospital discharge
Population: Number of participants analyzed represent those enrolled and randomized minus those withdrawn or lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 69 | 76
Participants | 55 | 71
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.03, Fisher Exact

6. Secondary Outcome: Correct Medication Frequency
Description: Participants (caregivers) will be asked in a follow-up survey to provide the frequency of their child's discharge medication. This will be scored as correct if it matches the frequency of the medication prescribed in the electronic health record.
Time Frame: During follow-up survey assessment 48-72 hours following hospital discharge
Population: Number of participants analyzed represent those enrolled and randomized minus those withdrawn or lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 69 | 76
Participants | 65 | 74
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.42, Fisher Exact

7. Other Pre Specified Outcome: Correct Medication Duration
Description: Participants (caregivers) will be asked in a follow-up survey to provide the total duration of their child's discharge medication. This will be scored as correct if it matches the duration of the medication prescribed in the electronic health record.
Time Frame: During follow-up survey assessment 48-72 hours following hospital discharge
Population: Number of participants analyzed represent those enrolled and randomized minus those withdrawn or lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 69 | 76
Participants | 49 | 65
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.04, Fisher Exact

8. Other Pre Specified Outcome: Correct Medication Side Effects
Description: Participants (caregivers) will be asked in a follow-up survey to provide the medication side effects of their child's discharge medication. Caregivers will receive 1 point for every correctly identified side effect as it matches a list of pre-specified side effects determined by the study team. Caregivers will receive no points if they are unable to name any side effects on the prespecified list.
Time Frame: During follow-up survey assessment 48-72 hours following hospital discharge
Population: Number of participants analyzed represent those enrolled and randomized minus those withdrawn or lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 69 | 76
Participants | 13 | 60
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p < 0.001, Fisher Exact

9. Other Pre Specified Outcome: Correct Medication Storage
Description: Participants (caregivers) will be asked in a follow-up survey to provide the correct recommended storage location of their child's discharge medication. This will be scored as correct if it matches the recommended storage location of the medication prescribed in the electronic health record.
Time Frame: During follow-up survey assessment 48-72 hours following hospital discharge
Population: Number of participants analyzed represent those enrolled and randomized minus those withdrawn or lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 69 | 76
Participants | 67 | 76
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.22, Fisher Exact

ADVERSE EVENTS:
Description: Death, serious adverse events, and nonserious adverse events were not assessed for study participants as this was a minimal-risk, behavioral intervention.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT05143047/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT05143047/ICF_000.pdf